CLINICAL TRIAL: NCT03093662
Title: Analysis of Preoxygenation Combining Nasal Cannula With Noninvasive Positive Pressure Ventilation: A Randomized Crossover Trial
Brief Title: Preoxygenation With Nasal Cannula and Noninvasive Positive Pressure Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Program Director for Research, Emergency Medicine, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: C.2017.011
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Cannula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ventilation with nasal cannula (Experimental): Non-invasive positive pressure ventilation with nasal cannula.
  Interventions: Device: Ventilation with nasal cannula; Device: Ventilation without nasal cannula
- Ventilation without nasal cannula (Active Comparator): Non-invasive positive pressure ventilation without nasal cannula.
  Interventions: Device: Ventilation with nasal cannula; Device: Ventilation without nasal cannula

INTERVENTIONS:
Device: Ventilation with nasal cannula — Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear) while simultaneously wearing nasal cannula (Carefusion AirLife Standard Nasal Cannula) with 15 L/min oxygen flow. Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
Device: Ventilation without nasal cannula — Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear). Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).

SUMMARY:
This is a prospective randomized cross over study of healthy volunteers comparing end-tidal oxygen concentration among subjects undergoing continuous positive airway pressure ventilation via a noninvasive ventilation (NIV) mask with and without the addition of nasal cannulas.

DETAILED DESCRIPTION:
Noninvasive positive pressure ventilation with the addition of a nasal cannula is a useful technique to pre-oxygenate and provide apneic oxygenation in hypoxic patients undergoing emergency airway management. This study aims to evaluate preoxygenation by quantifying end-tidal oxygen (etO2) concentration resulting from nasal cannula placement underneath a noninvasive positive pressure ventilation (NIPPV) mask. This is a prospective randomized cross over study of healthy volunteers undergoing continuous positive airway pressure ventilation via a noninvasive ventilation (NIV) mask with and without the addition of nasal cannulas. End-tidal oxygen concentration will be measured by an oxygen sensor following three minutes of NIPPV with and without the addition of a nasal cannula, with each subject serving as his or her own control.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy volunteer aged 18-65 years.

Exclusion Criteria:

* Previous inability to tolerate noninvasive positive pressure ventilation with addition of a nasal cannula.
* Known underlying cardiac or pulmonary disease.
* Active respiratory infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Brown, MD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Background] Sakles JC, Mosier JM, Patanwala AE, Arcaris B, Dicken JM. First Pass Success Without Hypoxemia Is Increased With the Use of Apneic Oxygenation During Rapid Sequence Intubation in the Emergency Department. Acad Emerg Med. 2016 Jun;23(6):703-10. doi: 10.1111/acem.12931. Epub 2016 May 13. PMID 26836712
- [Background] Bodily JB, Webb HR, Weiss SJ, Braude DA. Incidence and Duration of Continuously Measured Oxygen Desaturation During Emergency Department Intubation. Ann Emerg Med. 2016 Mar;67(3):389-95. doi: 10.1016/j.annemergmed.2015.06.006. Epub 2015 Jul 9. PMID 26164643
- [Background] Hayes-Bradley C, Lewis A, Burns B, Miller M. Efficacy of Nasal Cannula Oxygen as a Preoxygenation Adjunct in Emergency Airway Management. Ann Emerg Med. 2016 Aug;68(2):174-80. doi: 10.1016/j.annemergmed.2015.11.012. Epub 2015 Dec 31. PMID 26747218

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventilation With Nasal Cannula First, Then Without Nasal Cannula: First intervention: subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear) while simultaneously wearing nasal cannula (Carefusion AirLife Standard Nasal Cannula) with 15 L/min oxygen flow. Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
  Second intervention: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear). Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
- Ventilation Without Nasal Cannula First, Then With Nasal Cannula: First intervention: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear). Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
  Second intervention: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear) while simultaneously wearing nasal cannula (Carefusion AirLife Standard Nasal Cannula) with 15 L/min oxygen flow. Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
Period: First Intervention (3 Minutes)
Arm/Group | Ventilation With Nasal Cannula First, Then Without Nasal Cannula | Ventilation Without Nasal Cannula First, Then With Nasal Cannula
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: Washout Period (5 Minutes)
Arm/Group | Ventilation With Nasal Cannula First, Then Without Nasal Cannula | Ventilation Without Nasal Cannula First, Then With Nasal Cannula
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: Second Intervention (3 Minutes)
Arm/Group | Ventilation With Nasal Cannula First, Then Without Nasal Cannula | Ventilation Without Nasal Cannula First, Then With Nasal Cannula
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ventilation With Nasal Cannula First: Non-invasive positive pressure ventilation with nasal cannula first followed by non-invasive positive pressure ventilation without nasal cannula.
  Ventilation with nasal cannula: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear) while simultaneously wearing nasal cannula (Carefusion AirLife Standard Nasal Cannula) with 15 L/min oxygen flow. Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
  Ventilation without nasal cannula: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear). Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
- Ventilation Without Nasal Cannula First: Non-invasive positive pressure ventilation without nasal cannula first followed by non-invasive positive pressure ventilation with nasal cannula.
  Ventilation with nasal cannula: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear) while simultaneously wearing nasal cannula (Carefusion AirLife Standard Nasal Cannula) with 15 L/min oxygen flow. Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
  Ventilation without nasal cannula: Subject is fitted with a face mask and undergoes three continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear). Subject then removes mask and immediately exhales into an oxygen sensor (Maxtec Max-250E).
- Total: Total of all reporting groups
Arm/Group | Ventilation With Nasal Cannula First | Ventilation Without Nasal Cannula First | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 13 | 13 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: End-tidal Oxygen
Description: Measured by exhalation into sensor (Maxtec Max-250E)
Time Frame: 3 minutes after study start
Population: This was a cross-over study so ultimately all patients underwent both ventilation with nasal cannula and ventilation without nasal cannula; 18 underwent ventilation with nasal cannula first whereas the remaining 19 participants underwent ventilation without nasal cannula first. This design accounts for any combining of patients in analysis.
Measure: Mean (95% Confidence Interval); unit: End tidal oxygen saturation percentage
Arm/Group | Ventilation With Nasal Cannula | Ventilation Without Nasal Cannula
Number analyzed (Participants) | 37 | 37
End tidal oxygen saturation percentage | 78.1 [75.5 to 80.8] | 78.6 [75.6 to 81.4]

ADVERSE EVENTS:
Time Frame: Study duration (approximately 30 minutes).
Groups:
- Ventilation With Nasal Cannula: Subject is fitted with a face mask and undergoes 3 continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear) while simultaneously wearing nasal cannula (Carefusion AirLife Standard Nasal Cannula) with 15 L/min oxygen flow. Subject then removes mask and exhales into an oxygen sensor (Maxtec Max-250E).
  The cross over design means all patients eventually underwent both ventilation with nasal cannula and ventilation without nasal cannula, accounting for any combining of patients in analysis.
- Ventilation Without Nasal Cannula: Subject is fitted with a face mask and undergoes 3 continuous minutes of positive pressure ventilation (Respironics AF521, EE with CapStrap headgear). Subject then removes mask and exhales into an oxygen sensor (Maxtec Max-250E).
  The cross over design means all patients eventually underwent both ventilation with nasal cannula and ventilation without nasal cannula, accounting for any combining of patients in analysis.
Arm/Group | Ventilation With Nasal Cannula | Ventilation Without Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03093662/Prot_SAP_000.pdf